CLINICAL TRIAL: NCT02722850
Title: A Lifestyle Intervention Via Email (ALIVE) for Cancer Survivors
Brief Title: Web-based Study for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: M.D. Anderson Cancer Center (Other); The University of Texas Health Science Center, Houston (Other); University of Houston (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Raheem Paxton, Assistant Professor, University of North Texas Health Science Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 001
Record Dates: First submitted 2016-03-20; First posted 2016-03-30 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Physical Activity; Dietary Modification
Keywords: breast cancer; cancer survivorship; dietary intake; physical activity; quality of life
MeSH Terms: conditions — Motor Activity; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALIVE - Physical Activity (Experimental): PA CONDITION: The goal of the PA condition is to encourage participants to gradually increase moderate to vigorous PA to 150 minutes per week and to increase resistance training to a total of 15 minutes per day twice per week.
  Interventions: Behavioral: ALIVE
- ALIVE - Dietary Modification (Experimental): DIET CONDITION: The goal of the dietary condition includes increasing intake of fruit and vegetable to 5-servings per day. The program also encourages participants to increase the consumption of colorful fruits and vegetables. The fat goals consist of reducing saturated fats to <10% of total kilocalories per day, trans fats to <3 grams per day, and added sugar to <50 grams per day.
  Interventions: Behavioral: ALIVE

INTERVENTIONS:
Behavioral: ALIVE — ALIVE is an email-based platform designed to help participants increase their physical activity, increase fruit and vegetable consumption, and decrease their intake of saturated and trans fats and added sugars. This automated system contains content and tailoring that is delivered in the form of emails obtained directly from cancer patients. Additional information they will receive included: tips for achieving those goals, health information, and opportunities for interaction and engagement.

SUMMARY:
In this parallel group study, participants were randomized to either 1 of 3 conditions (a) fruit and vegetable consumption, (b) dietary fat and added sugars, or (c) physical activity.

DETAILED DESCRIPTION:
In this study, the investigators will evaluate the feasibility and preliminary results of a 3-month web-based lifestyle intervention 500 female cancer survivors.

Specific aim 1: to determine the rates of recruitment, retention, attendance, satisfaction, adverse events, and barriers to participation in the proposed intervention.

Specific aim 2: to determine whether a home-based intervention is associated with greater improvements in mean minutes of moderate to vigorous physical activity, diet quality, body size, constructs of Social Cognitive Theory, and health-related quality of life than participants randomized to a sedentary behavior reduction condition.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with breast cancer;
* 18-80 years old at time of cancer diagnosis;
* English-Speaking;
* Have access to high-speed internet.

Exclusion Criteria:

* Be currently enrolled in another intervention study or recently completed a study promoting healthy lifestyle behaviors (diet and/or exercise).
* Participants answering 'Yes' to one or more of the questions on the physical activity readiness questionnaire (PAR-Q) will need to obtain approval from a physician before they can participate in the intervention.
* Pregnant women will be excluded from the protocol.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Mean metabolic equivalent minutes of physical activity | 3-months
  Physical activity and sedentary behavior were assessed with the Work and Home Activity Questionnaire at baseline and at 3-months
Diet Quality | 3-month
  Dietary intake was assessed with Block health habits and history questionnaire. This instrument is a validated food frequency questionnaire

SECONDARY OUTCOMES:
Mean health related quality of life scores | 3-months
  Health-related quality of life will be assessed with instruments measuring functional status, pain and fatigue interference, and cognitive function at baseline and at 3-months.

CONTACTS AND LOCATIONS:
Overall Officials: Raheem Paxton, PhD, Principal Investigator — UNT - Health Science Center

IPD SHARING:
Plan to Share IPD: Undecided
Once data are compiled, the investigators will decide whether it will be available for sharing

REFERENCES:
- [Background] Sternfeld B, Block C, Quesenberry CP Jr, Block TJ, Husson G, Norris JC, Nelson M, Block G. Improving diet and physical activity with ALIVE: a worksite randomized trial. Am J Prev Med. 2009 Jun;36(6):475-83. doi: 10.1016/j.amepre.2009.01.036. PMID 19460655
- [Derived] Paxton RJ, Hajek R, Newcomb P, Dobhal M, Borra S, Taylor WC, Parra-Medina D, Chang S, Courneya KS, Block G, Block T, Jones LA. A Lifestyle Intervention via Email in Minority Breast Cancer Survivors: Randomized Parallel-Group Feasibility Study. JMIR Cancer. 2017 Sep 21;3(2):e13. doi: 10.2196/cancer.7495. PMID 28935620